CLINICAL TRIAL: NCT03612752
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effects of a Peptide-protein Extract (CMI-168) on Cognitive Function in Healthy Middle-aged Men and Women
Brief Title: CMI-168 on Cognitive Function in Healthy Middle-aged Men and Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cerebos Pacific Limited (Industry)
Responsible Party: Principal Investigator, Chaurjongh Hu, Professor, Cerebos Pacific Limited
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: N201711060
Record Dates: First submitted 2018-06-27; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Cognitive Change
Keywords: Chicken essence, cognitive function

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arm (Experimental): CMI-168
  Interventions: Dietary Supplement: CMI-168
- Placebo arm (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: CMI-168 — Dietary supplement
  Arms: Active arm
Other: Placebo — Placebo
  Arms: Placebo arm

SUMMARY:
The investigators propose to conduct the present study in order to primarily assess the effects of CMI-168 in neurocognition enhancement. Studies have shown that episodic memory performance is declined in elder populations showing elevated cortisol levels and cognitive decline is accelerated with greater levels of self-reporting perceived stress . Additionally, stress-related disorders such as depression and anxiety adversely affect and impair cognitive function. Given the significant role of chronic stress, sleep, depression and anxiety in impairing memory and learning performance, questionnaires used to measure the following parameters of stress (Perceived Stress Scale, PSS), sleep (Pittsburg Sleep Quality Index, PSQI), anxiety (State-Trait Anxiety Inventory, STAI) and depression (Beck Depression Inventory, BDI) have been incorporated into this study design. Additionally, levels of Brain-Derived Neurotrophic Factor (BDNF), a protein involved in neuronal survival and synaptic plasticity of the central and peripheral nervous system, have been reported to be significantly different in patients with depression or neurological disorders . The investigators will also examine the physiological levels of cortisol and BDNF in these subjects to determine their effect of CMI-168 supplementation on these measures, as well as the implications on cognition.

DETAILED DESCRIPTION:
Study participation will last approximately 14 weeks, comprising of up to 4 weeks for screening, 8 weeks-blinded supplementation period and 2 weeks post-supplementation period. During the 8 weeks period, subjects will take either 2 study tablets of CMI-168 or 2 tablets of matching placebo once daily in the morning. Supplementation will be stopped after 56 days and after another 14 days, subjects will be re-assessed.

Key assessment of the screening period will be the cognitive testing using the Cambridge Neuropsychological Test Automated Battery (CANTAB) to ensure that the subjects fall within the normal cognitive range for their ages. The study aims to only include subjects with normal cognition and showing no perceptible signs of cognitive impairment at screening (Visit 1). Subjects showing cognition abnormal cognition scores during the screening stage by the CANTAB assessment will not be included in the next stages of the study. After a screening period of 3 to 28 days, eligible subjects will be randomized 1:1 ratio to two treatment arms.

* CMI-168 (2 tablet, once daily, 56 days).
* Placebo (2 tablets once daily, 56 days)

Following randomisation,the various assessments including cognitive tests, questionnaires, event related potential and blood samples will be administered or taken at Visit 2 (Baseline, start of supplementation), Visit 3 (Day 28 supplementation) and Visit 4 (Day 56 supplementation) and Visit 5 (Day 70-2 weeks after termination of supplementation). Subject completion of the study will be defined as completing the assessments at Visit 5. The different tests will be administered according to the schedule of assessments below.

ELIGIBILITY:
Inclusion Criteria:

* Institutional Review Board approved written informed consent and privacy language as per national regulations must be obtained from the patient or legally authorized representative prior to any clinical study-related procedures
* Subject is an otherwise healthy male/female between 35-65 years of age during the study period.
* Patient has a body mass index range of 18.0 to 40.0 kg/m2, inclusive, and weighs at least 40 kg at screening
* Patient agrees not to participate in another interventional study while participating in the present study, defined as signing the informed consent form until completion of the study.
* Ability to understand and write Taiwanese Traditional Chinese or at least have completed Taiwan high school education
* Perceived Stress Scale Score> 20
* Within normal cognition range as assessed by CANTAB battery

Exclusion Criteria:

* Inability to participate in the evaluation of the study
* Subject is pregnant at the time of the screening assessment
* Active viral infection or bacterial infection based on clinical observations
* Visual or hearing impairment sufficient to preclude cooperation with neurocognitive testing
* Long-term consumption of dietary supplement or herbal products likely to have an effect on memory
* Subjects intolerant or allergic to protein-based food or supplement
* Subjects with significant cognitive impairment including already being diagnosed with Alzheimer's disease, Parkinson's disease, schizophrenia or dementia.
* History of cardiovascular disease, respiratory disease, head injury, cancer, diabetes or neuropsychological disease
* Life threatening pathology (such as cancer) in remission for less than 1 year or still ongoing
* Psychological or linguistic incapability to sign the informed consent
* Anti-depressant treatment stopped since less than 3 months or still ongoing
* History of allergy to chicken meat
* Pregnant or lactating women
* Smoking more than 10 cigarettes per day
* Suspected or known alcohol abuse or addiction
* Subjects with any other conditions or diseases that investigator consider as not appropriate to be entered in the study

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Change of Cognitive function | From Day 0 to Day 28, Day 56 and Day 70
  Cambridge Neuropsychological Test Automated Battery (CANTAB)
Change of Word Lists Subtest of the Weschler Memory Scale 3rd edition | From Day 0 to Day 28, Day 56 and Day 70
  Word Lists Subtest of the Weschler Memory Scale 3rd edition
Change of Logical Memory Subtest of Weschler Memory Scale 3rd edition | From Day 0 to Day 28, Day 56 and Day 70
  Logical Memory Subtest of Weschler Memory Scale 3rd edition
Change of Family Pictures Subtest of Weschler Memory Scale 3rd edition | From Day 0 to Day 28, Day 56 and Day 70
  Family Pictures Subtest of Weschler Memory Scale 3rd edition

SECONDARY OUTCOMES:
Change of serum ALT | From Day 0 to Day 28, Day 56 and Day 70
  serum ALT
Change of serum AST | From Day 0 to Day 28, Day 56 and Day 70
  serum AST
Change of serum BUN | From Day 0 to Day 28, Day 56 and Day 70
  serum BUN
Change of serum creatinin | From Day 0 to Day 28, Day 56 and Day 70
  serum creatinin
Change of serum T3 | From Day 0 to Day 28, Day 56 and Day 70
  serum T3
Change of serum T4 | From Day 0 to Day 28, Day 56 and Day 70
  serum T4
Change of serum TSH | From Day 0 to Day 28, Day 56 and Day 70
  serum TSH
Change of serum cortisol at 8 am | From Day 0 to Day 28, Day 56 and Day 70
  serum cortisol at 8 am
Change of serum fasting sugar | From Day 0 to Day 28, Day 56 and Day 70
  serum fasting sugar
Change of Event related potential P300 | From Day 0 to Day 28, Day 56 and Day 70
  Event related potential P300
Change of Perceived Stress Scale (PSS) | From Day 0 to Day 28, Day 56 and Day 70
  Perceived Stress Scale (PSS)
Change of State-Trait Anxiety Inventory (STAI) | From Day 0 to Day 28, Day 56 and Day 70
  State-Trait Anxiety Inventory (STAI)
Change of Beck Depression Inventory (BDI) | From Day 0 to Day 28, Day 56 and Day 70
  Beck Depression Inventory (BDI)
Change of Pittsburgh Sleep Quality Index (PSQI) | From Day 0 to Day 28, Day 56 and Day 70
  Pittsburgh Sleep Quality Index (PSQI)
Change of serun brain-derived neurotrophic factor (BDNF) | From Day 0 to Day 28, Day 56 and Day 70
  serum brain-derived neurotrophic factor (BDNF)

CONTACTS AND LOCATIONS:
Overall Officials: Chaurjong Hu, MD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University - Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu D, Yang CC, Chen KY, Lin YC, Wu PJ, Hsieh PH, Nakao Y, Ow MYL, Hsieh YC, Hu CJ. Hydrolyzed Chicken Extract (ProBeptigen(R)) on Cognitive Function in Healthy Middle-Aged People: A Randomized Double-Blind Trial. Nutrients. 2020 May 10;12(5):1362. doi: 10.3390/nu12051362. PMID 32397609